CLINICAL TRIAL: NCT01219543
Title: A Phase I, Open-label, Multicentre, Dose Escalation Study to Assess the Safety and Tolerability, and Pharmacokinetics of AZD1480 in Asian Patients With Advanced Solid Malignancies and Asian Patients With Child-Pugh A to B7 Advanced Hepatocellular Carcinoma (HCC) in the Escalation Phase, Estimated Glomerular Filtration Rate(EGFR) or ROS Mutant NSCLC and Non-smokers With Lung Metastasis and Gastric Cancer and Solid Tumour With Biopsy Available in the Expansion Phase.
Brief Title: A Phase I Study of AZD1480 in Patients With Advanced Solid Malignancies and Advanced Hepatocellular Carcinoma in the Escalation Phase,Non-Small Cell Lung Cancer(NSCLC) and Non-smokers With Lung Metastasis and Gastric Cancer and Solid Tumour in the Expansion Phase.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Compound development discontinued
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1060C00004
Record Dates: First submitted 2010-10-11; First posted 2010-10-13 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Solid Tumour; Advanced Solid Malignancies; Child-Pugh A to B7 Advanced Hepatocellular Carcinoma; EGFR and/or ROS Mutant NSCLC; Lung Metastasis Carcinoma; Gastric Cancer
Keywords: Advanced solid malignancies; Child-Pugh A to B7 advanced hepatocellular carcinoma; EGFR and/or ROS mutant NSCLC; Non-smokers with lung metastasis; Gastric cancer; Solid tumour; AZD1480; JAK1/JAK2 kinase inhibitor
MeSH Terms: conditions — Stomach Neoplasms

ARMS (4):
- Part A (Experimental): Daily dosing of AZD1480 to the patients with solid tumours excluding HCC
  Interventions: Drug: AZD1480 Daily
- Part B (Experimental): BID dosing of AZD1480 to the patients with advanced HCC (Child-Pugh A to B7)
  Interventions: Drug: AZD1480 BID
- Part C (Experimental): BID dosing of AZD1480 to the patients with solid tumours excluding HCC
  Interventions: Drug: AZD1480 BID
- Expansion (Experimental): BID dosing of AZD1480 to the patients with EGFR or ROS mutant NSCLC and non-smokers with lung metastasis and gastric cancer and solid tumour with biopsy available.
  Interventions: Drug: AZD1480 BID

INTERVENTIONS:
Drug: AZD1480 Daily — Oral Dose, Capsule, Daily Dosing
  Arms: Part A
Drug: AZD1480 BID — Oral Dose, Capsule, BID Dosing
  Arms: Expansion; Part B; Part C

SUMMARY:
This is Phase I, open-label and dose escalation study to evaluate the safety and tolerability of AZD1480(JAK2 inhibitor) in Asian patients with advanced solid tumors (Part A and C) and in patients with advanced HCC (Part B) in the escalation phase, EGFR or ROS mutant NSCLC and non-smokers with lung metastasis and gastric cancer in the expansion phase and to evaluate daily and BID dosing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older
* For Part A and C: Histological or cytological confirmation of a solid malignant tumour refractory to standard therapies or for which no standard therapies exist. Patients with lymphoma & HCC are excluded.
* For Expansion : Histological or cytological confirmation of
* Expansion 1: EGFR and/or ROS mutant NSCLC or Non-smokers with lung metastasis
* Expansion 2: Gastric cancer or solid tumour with biopsy available (consenting paired biopsies)refractory to standard therapies or for which no standard therapies exist. Patients with lymphoma & HCC are excluded.
* For Part B : Advanced or metastatic HCC, unresectable and incurable with ablative therapy or TACE, with no standard therapy available.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 with no deterioration over the previous 2 weeks
* For Part B : Child-Pugh liver function status classified as A to B7

Exclusion Criteria:

* For any other chemotherapy, immunotherapy or anticancer agents, within 5 half lives or 3 weeks must have elapsed from treatment to of the first dose of investigational product, whichever is shorter.
* With the exception of alopecia, any unresolved toxicities from prior therapy ≥ Grade 2 of CTCAE V4.02 at the time of starting study (except LFTs for HCC patients, which may be Grade 2 at the time of starting the study)
* Any of the following conditions:Interferon treatment for HBV and HCV Prior Liver Transplantation
* Inadequate bone marrow reserve or organ function as demonstrated by laboratory values
* Evidence of established interstitial lung disease(ILD) on baseline high resolution computerized tomography(HRCT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To investigate the safety and tolerability of AZD1480 | Safety and tolerability monitoring will proceed for whole study period. Screening, Cycle1Day1, Cycle1Day5 (only for Part B), Cycle1Day8, Cycle1Day15, Cycle2Day1, Cycle2Day8 and Day1 of further Cycles, IP discontinued visit and 30-days follow up

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics (PK) of AZD1480 following single dose and multiple doses | Part A and Expansion - 12 times during Cycle 1, 11 times during Cycle 2. Part B and C - 11 times during Cycle 1, 10 times during Cycle 2. *1 additional PK sample in Cycle 1 will be collect for optional biopsy sample collected patients.
To obtain a preliminary assessment of the anti-tumour activity of AZD1480 | Tumour response assessment by RECIST (Response Evaluation Criteria In Solid Tumors) version 1.1 every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Becker Hewes, MD, Study Director — AstraZeneca; Kang Yoon-Koo, MD, PhD, Principal Investigator — Asian Medical Center
Locations (1):
- Research Site, Seoul, South Korea